CLINICAL TRIAL: NCT00284375
Title: Systematic Registration of All Big Toe Prostheses Placed in Ghent University Hospital
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2005/016
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Big Toe Prosthesis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Registration of all big toe prostheses in Ghent University Hospital — Registration of all big toe prostheses in Ghent University Hospital.

SUMMARY:
Systematic registration of all big toe prostheses placed in Ghent University Hospital for analyses of global results, comparison between different types of prostheses, ...

ELIGIBILITY:
Inclusion Criteria:

* Big toe prosthesis

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 500 patients will be included.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frequency of big toe prostheses. | ongoing basis
  Developing a database of all big toe prostheses in Ghent University Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Bongaerts, MD, Principal Investigator — University Hospital, Ghent; Jeroen De Vil, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be